CLINICAL TRIAL: NCT06916416
Title: Phase II Trial of Anti-PD-1 Antibody Treatment and Radiotherapy in Early-stage Favorable Classic Hodgkin Lymphoma
Acronym: PREFer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Dr. Dennis Eichenauer, Dr., University of Cologne
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Uni-Koeln-5450; 2024-520138-31-00 (EU CTIS Number)
Record Dates: First submitted 2025-03-31; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Classical Hodgkin Lymphoma
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab (Experimental): All patients will receive 6 doses of 200mg Pembrolizumab iv as single agent every three weeks followed by 20Gy radiotherapy
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — 6 doses of 200mg Pembrolizumab iv as single agent every three weeks followed by radiotherapy 20Gy

SUMMARY:
By the implementation of the anti-PD-1 antibody pembrolizumab and given its possible synergy with RT, the aim of the present trial is to develop a chemotherapy-free first-line treatment for patients with newly diagnosed early-stage favorable cHL.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven first diagnosis of cHL
* Stage I-II without risk factors

  * Large mediastinal mass
  * Extranodal involvement
  * Elevated erythrocyte sedimentation rate (ESR)
  * Involvement of ≥ 3 nodal areas

Exclusion Criteria:

* Central nervous system lymphoma, nodular lymphocyte-predominant Hodgkin lymphoma or composite lymphoma,
* Prior cHL-directed treatment
* Prior chemotherapy, RT or allogeneic stem cell/solid organ transplant
* Prior or concurrent disease precluding protocol treatment (for details see section 4.2)
* Pregnancy or breastfeeding
* Non-compliance

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | PFS at 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Eichenauer, Dr., Principal Investigator — University Hospital of Cologne

IPD SHARING:
Plan to Share IPD: Undecided